CLINICAL TRIAL: NCT06869993
Title: Food and Families: a Pilot Study of the Acceptability, Feasibility, and Mental Health Effects of a Meal Kit Intervention in Rural, Low-Income Families
Brief Title: Giving Healthy Meal Kits and Cooking Lessons to Rural Families with Food Insecurity.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Lauren Ciszak, Postdoctoral Fellow, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Food and Families; 2268160-1 (Other Grant/Funding Number: MaineHealth)
Record Dates: First submitted 2025-03-02; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Food Insecurity; Food Insecurity Among Children; Social Emotional Wellness; Caregiver Stress; Caregiver Distress; Caregiver Mental Health; Family Function; Family Functioning; Nutrition; Child Mental Health
Keywords: Food is Medicine; Family Stress; Child stress; Food Insecurity; Childhood Food Insecurity; Child Mental Health; Nutrition; family; Family Functioning; Mental Health; Caregiver Stress; Child Caregiver; Healthy Food; Nutrition Security; Nutrition Insecurity
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): Participants will receive 4 weeks of health meal kits delivered to their homes in addition culinary medicine education via an app. They will also participate in weekly as well as pre-and post-intervention assessments.
  Interventions: Dietary Supplement: Meal Kit plus Mobile Culinary Medicine Education

INTERVENTIONS:
Dietary Supplement: Meal Kit plus Mobile Culinary Medicine Education — This intervention will involve four phases: (1) a baseline assessment; (2) a 7-day monitoring phase, (3) a 30-day intervention phase in which all households receive weekly meal kits delivered to their home in addition to mobile culinary medicine education; and (4) a follow-up assessment.

SUMMARY:
The goal of this clinical trial is to learn if providing healthy meal kits to food insecure families can help lessen the social and emotional impacts of food insecurity on kids and their caregivers in rural Maine. The main questions it aims to answer are:

1. Is receiving healthy meal kits delivered to homes feasible and acceptable to rural Maine families?
2. Does receiving meal kits (along with an app to help learn how to cook the food) improve food insecurity and diet quality in rural Maine families?
3. Does receiving meal kits (along with an app to help learn how to cook the food) improve family function in rural Maine families? We will look at caregivers' stress, family conflict, household chaos, and child emotional-behavioral symptoms.

Participants will:

1. Recieve and prepare a dietitian-designed meal kit with 10 meals per week for 4 weeks.
2. Receive free culinary medicine education via an app that they will continue to have access to after the study ends.
3. Complete a 1-1.5 hour virtual visit at the beginning of and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Legal caregiver for a child between the ages of 6-12 with whom they live at least 75% of the time.
* Reside in rural county in Maine as designated by the Health Resources and Services Administration.
* Endorse food insufficiency within the past month on their screening questionnaire.
* Able to speak and read in English.
* Stable address with the ability to receive packages

Exclusion Criteria:

* Inadequate access (<5 days/week) to a kitchen with refrigeration and heating elements to prepare meals.
* Food-restrictive diet (i.e., veganism, gluten-free, dialysis-dependent, severe heart failure).
* A household member with any anaphylactic food allergy.
* No access to a smartphone with texting capabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
USDA Household Food Security Survey | Baseline and 5 weeks
  An 18-item questionnaire designed to assess a household's level of food insecurity during the past year, including questions related to both worry and insufficiency in relation to both adults and children living in the household
Rapid Prime Diet Quality Screener | Baseline and 5 weeks
  A 13-item diet screener that assesses the frequency with which various categories of food were consumed over the past month (e.g., processed meats, vegetables, soft drinks).
Confusion, Hubbub, and Order Scale | Baseline and 5 weeks
  A 15-item, caregiver-report questionnaire that assesses the level of environmental confusion in the home
24-Hour Food Recall | Baseline and 5 weeks
  A structured assessment intended to capture detailed information about all foods, beverages, and dietary supplements consumed by the participant in the past 24 hours. The assessment queries about the time of day, portion size, and preparation methods of each food item.
Cooking and Food Provisioning Action Scale | Baseline and 5 weeks
  A 28-question validated questionnaire assessing food agency in three separate categories (self-efficacy, structure, and attitude).
Parenting Stress Index - Short Form | Baseline and 5 weeks
  A 36-item caregiver report assesses three domains of stress (parental distress, dysfunctional parent-child interactions, and difficult child).
Perceived Stress Scale | Baseline and 5 weeks
  A 10-item, self-report measure that assesses the degree to which different situations are appraised as stressful, unpredictable, and uncontrollable.
Alabama Parenting Questionnaire - Short Form | Baseline and 5 weeks
  A 9-item, caregiver-report measure of parenting practices that assesses domains of positive parenting, poor monitoring/supervision, and inconsistent discipline
Family Environment Scale - Fourth Edition | Baseline and 5 weeks
  A self-report assessment designed to assess different aspects of family functioning via 90 true or false questions. In order to reduce participant burden, only items from the Cohesion, Conflict, Organization and Control subscale will be administered.
Child Behavior Checklist | Baseline and 5 weeks
  The Child Behavior Checklist (CBCL) is a caregiver-report measure that consist of 120 problem items rated on a three-point scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true) that yield empirically derived subscales related to different psychological symptoms and competence in several areas of functioning. Subscales are consistent across age, gender, informant, and culture and have test-retest reliabilities between 0.74 and 0.95 and Cronbach alphas between 0.79 and 0.97. The Brief Problem Monitor is a 19-item caregiver-report measure with parallel items and scales to the CBCL designed for assessing change over time.

SECONDARY OUTCOMES:
Adult Self-Report | Baseline and 5 weeks
  A self-report inventory on which caregivers rated the extent to which they have experienced 126 psychological problems during the past six months on a three-point scale 1 = somewhat or sometimes true, 2 = very true or often true). Items form empirically validated subscales that are normed by age, gender, and culture.
PROMIS Fatigue Profile | Baseline and 5 weeks
  16-item, self-report measure that assesses fatigue intensity and its effects on social functioning, cognition, and motivation.
Positive and Negative Affect Schedule | Baseline and 5 weeks
  A 20-item self-report measure that assesses the extent to which participants have various moods during a specified timeframe (i.e., 30 days) which yields independent positive and negative affect subscales.

OTHER OUTCOMES:
Demographic Survey | Baseline
  A 14-item questionnaire designed specifically for the current study was used to obtain basic information about the caregiver (e.g., age, gender identity, race, ethnicity, occupation, and level of education) as well as the composition and economic circumstances of the household.

CONTACTS AND LOCATIONS:
Overall Officials: Merelise Ametti, PhD, MPH, Principal Investigator — MaineHealth; Lauren Ciszak, MD, Principal Investigator — MaineHealth
Locations (1):
- MaineHealth, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No
For patient protection IPD will not be shared.